CLINICAL TRIAL: NCT01705691
Title: A Phase II Randomized Clinical Trial Evaluating Neoadjuvant Chemotherapy Regimens With Weekly Paclitaxel or Eribulin Followed by Doxorubicin and Cyclophosphamide in Women With Locally Advanced HER2-Negative Breast Cancer
Brief Title: Comparison of Neoadjuvant Chemotherapy With Weekly Paclitaxel or Eribulin Followed by A/C in Women With Locally Advanced HER2-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-9
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; eribulin; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Paclitaxel then AC (Active Comparator): Paclitaxel 80 mg/m2 IV weekly for 12 doses followed by doxorubicin and cyclophosphamide IV every 21 days for 4 cycles
  Interventions: Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm 2: Eribulin then AC (Experimental): Eribulin 1.4 mg/m2 IV on days 1 and 8 of a 21-day cycle for 4 cycles, followed by doxorubicin and cyclophosphamide IV every 21 days for 4 cycles
  Interventions: Drug: Eribulin; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Paclitaxel — 80 mg/m2 IV over 60 minutes weekly for 12 weeks
  Arms: Arm 1: Paclitaxel then AC
Drug: Eribulin — 1.4 mg/m2 IV over 2 to 5 minutes on Days 1 and 8 every 21 days for 4 cycles
  Other Names: eribulin mesylate
  Arms: Arm 2: Eribulin then AC
Drug: Doxorubicin — 60 mg/m2 IV over 15 minutes on day 1 every 21 days for 4 cycles
Drug: Cyclophosphamide — 600 mg/m2 IV over 30 minutes on day 1 every 21 days for 4 cycles

SUMMARY:
NSABP FB-9 is a Phase II, multi-center, randomized study of eribulin or weekly paclitaxel followed by doxorubicin and cyclophosphamide (AC) as neoadjuvant therapy for women with HER2-negative, operable and locally advanced breast cancer (stage IIb and III). Patients in the control arm will receive neoadjuvant weekly paclitaxel (WP) followed by AC. The primary aim of the study is to determine the pathologic complete response (ypCR) in breast and axillary lymph nodes following completion of neoadjuvant therapy. The secondary aims include determination of the ypCR in axillary nodes, clinical complete response (ycCR) rate after eribulin or paclitaxel and after completion of neoadjuvant chemotherapy, two-year recurrence-free interval, two-year overall survival, and toxicity of the neoadjuvant regimens.

DETAILED DESCRIPTION:
Patients will be randomized to one of two neoadjuvant therapy regimens. Patients in Arm 1 will receive WP 80 mg/m2 for 12 doses followed by standard AC every 21 days for 4 cycles. Patients in Arm 2 will receive 4 cycles of eribulin 1.4 mg/m2 on days 1 and 8 of a 21-day cycle followed by standard AC every 21 days for 4 cycles. As soon as possible following recovery from chemotherapy, the patient will have either lumpectomy or mastectomy and axillary staging.

In both arms, clinical response will be assessed by physical exam on day 1 of each study therapy cycle. MRI of the breast is required within 4 weeks prior to randomization and following completion of eribulin or WP (before starting AC). Following recovery from surgery, patients will receive radiation therapy and hormonal therapy as clinically indicated. Other postoperative therapies are prohibited.

Patients will be randomized to the control arm (Arm 1) and to the investigational arm (Arm 2) in a 1:2 ratio. The sample size will be up to 50 patients with about 30 patients in Arm 2 and about half that number in Arm 1. Accrual is expected to occur over 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a life expectancy of at least 10 years, excluding their diagnosis of breast cancer. (Comorbid conditions should be taken into consideration, but not the diagnosis of breast cancer.)
* Patients of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy and for at least 6 months after the last dose of study therapy.
* The patient must have consented to participate and must have signed and dated an appropriate Institutional Review Board (IRB)-approved consent form that conforms to federal and institutional guidelines.
* Patients must be female.
* Patients must be > 18 years old.
* The Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1.
* The diagnosis of invasive adenocarcinoma of the breast must have been made by core needle biopsy or by limited incisional biopsy.
* Patients must have ER analysis performed on the primary tumor prior to randomization. If ER analysis is negative, then Progesterone Receptor (PgR) analysis must also be performed. (Patients are eligible with either hormone receptor-positive or hormone receptor-negative tumors.)
* Clinical staging, based on the assessment by physical exam, must be American Joint Committee on Cancer (AJCC) stage IIB, IIIA, IIIB, or IIIC: cT2 and cN1, cT3 and cN0 or cN1, Any cT and cN2 or cN3, cT4
* The patient must have a mass in the breast or axilla measuring greater than or equal to 2.0 cm by physical exam, unless the patient has inflammatory breast cancer, in which case measurable disease by physical exam is not required.
* At the time of randomization, blood counts performed within 4 weeks prior to randomization must meet the following criteria: Absolute Neutrophil Count (ANC) must be greater than or equal to 1200/mm3; Platelet count must be greater than or equal to 100,000/mm3; Hemoglobin must be greater than or equal to 10 g/dL.
* The following criteria for evidence of adequate hepatic function performed within 4 weeks prior to randomization must be met: total bilirubin must be less than or equal to Upper Limit of Normal (ULN) for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and alkaline phosphatase must be less than or equal to 1.5 x ULN for the lab; and Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) must be less than or equal to 1.5 x ULN for the lab.
* Patients with alkaline phosphatase > ULN but less than or equal to 1.5 x ULN are eligible for inclusion in the study if liver imaging (CT, MRI, PET, or PET-CT scan) performed within 4 weeks prior to randomization does not demonstrate metastatic disease and the requirements in the criteria below for unexplained skeletal pain are met.
* Patients with either unexplained skeletal pain or alkaline phosphatase that is > ULN but less than or equal to 1.5 x ULN are eligible for inclusion in the study if a bone scan, PET-CT scan, or PET scan performed within 4 weeks prior to randomization does not demonstrate metastatic disease. Patients with suspicious findings on bone scan or PET scan are eligible if suspicious findings are determined to be benign by x-ray, MRI, or biopsy.
* Serum creatinine performed within 4 weeks prior to randomization must be less than or equal to 1.5 x ULN for the lab.
* Serum potassium and serum magnesium performed within 4 weeks prior to randomization must be Within Normal Limits (WNL).
* The Left Ventricular Ejection Fraction (LVEF) assessment by 2-D echocardiogram or Multigated acquisition (MUGA) scan performed within 90 days prior to randomization must be greater than or equal to 50% regardless of the facility's Lower Limit of Normal (LLN).
* ECG performed within 4 weeks before study entry must demonstrate a QTc interval that is less than or equal to 0.47 seconds.

Exclusion Criteria:

* Tumor that has been determined to be HER2-positive by immunohistochemistry (3+) or by in situ hybridization (positive for gene amplification), or has been determined to be HER2-equivocal and the investigator plans to administer trastuzumab or other targeted therapy.
* Fine Needle Aspiration (FNA) alone to diagnose the primary breast cancer.
* Excisional biopsy or lumpectomy performed prior to randomization.
* Surgical axillary staging procedure prior to randomization. (Procedures that are permitted prior to study entry include: 1) FNA or core biopsy of an axillary node for any patient, and 2) although not recommended, a pre-neoadjuvant therapy Sentinal Node (SN) biopsy for patients with clinically negative axillary nodes.)
* Definitive clinical or radiologic evidence of metastatic disease. (Note: Chest imaging is mandatory for all patients within 90 days prior to randomization. Other imaging [if required] must have been performed within 4 weeks prior to randomization.)
* History of ipsilateral invasive breast cancer regardless of treatment or ipsilateral Ductal Carcinoma in Situ (DCIS) treated with Radiation Therapy (RT). (Patients with a history of Lobular Carcinoma in Situ (LCIS), contralateral DCIS [regardless of RT], or contralateral invasive breast cancer are eligible.)
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior to randomization.
* Known metastatic disease from any malignancy (solid tumor or hematologic).
* Previous therapy with anthracyclines, taxanes, cyclophosphamide, or eribulin for any malignancy.
* Treatment including RT, chemotherapy, and/or targeted therapy, administered for the currently diagnosed breast cancer prior to randomization.
* Continued endocrine therapy such as raloxifene or tamoxifen (or other SERM) or an aromatase inhibitor. (Patients are eligible if these medications are discontinued prior to randomization.)
* Any continued sex hormonal therapy, e.g., birth control pills and ovarian hormone replacement therapy. Patients are eligible if these medications are discontinued prior to randomization.
* Requirement for chronic use of any drugs known to prolong the QT interval, including Na+ and K+ channel blockers. (Patients are eligible if these medications and/or substances can be discontinued prior to the first dose of eribulin and will not need to be resumed until after the last dose of eribulin.)
* Active hepatitis B or hepatitis C with abnormal liver function tests.
* Intrinsic lung disease resulting in dyspnea.
* Active infection; or chronic infection requiring chronic suppressive antibiotics.
* Persistent greater than or equal to grade 2 diarrhea regardless of etiology.
* Sensory or motor neuropathy greater than or equal to grade 2, as defined by the NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0.
* Conditions that would prohibit intermittent administration of corticosteroids for paclitaxel premedication.
* Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids).
* Uncontrolled hypertension defined as a systolic BP > 150 mmHg or diastolic BP > 90 mmHg, with or without anti-hypertensive medications. (Patients with hypertension that is well-controlled on medication are eligible.)
* Cardiac disease (history of and/or active disease) that would preclude the use of any of the drugs included in the treatment regimen. This includes but is not confined to: Active cardiac disease: symptomatic angina pectoris within the past 180 days that required the initiation of or increase in anti-anginal medication or other intervention; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; and symptomatic pericarditis. History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of Left Ventricular (LV) function; history of documented Congestive Heart Failure (CHF) documented cardiomyopathy; and congenital long QT syndrome.
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Pregnancy or lactation at the time of randomization.
* Any psychiatric or addictive disorder or other condition that, in the opinion of the investigator, would preclude her from meeting the study requirements.
* Use of any investigation agent within 4 weeks prior to randomization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (20):
- United States (18):
  - CCOP, Colorado Cancer Research Program, Inc., Denver, Colorado
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Henry Ford Health System, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Carolinas Medical Center/Levine Cancer Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital/Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - NSABP Foundation, Inc., Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
- Canada (2):
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Abraham J, Robidoux A, Tan AR, Limentani S, Sturtz K, Shalaby I, Alcorn H, Buyse ME, Wolmark N, Jacobs SA. Phase II randomized clinical trial evaluating neoadjuvant chemotherapy regimens with weekly paclitaxel or eribulin followed by doxorubicin and cyclophosphamide in women with locally advanced HER2-negative breast cancer: NSABP Foundation Study FB-9. Breast Cancer Res Treat. 2015 Jul;152(2):399-405. doi: 10.1007/s10549-015-3466-4. Epub 2015 Jul 1. PMID 26126970

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient randomly assigned to Arm 2 withdrew consent before receiving protocol therapy.
Period: Overall Study
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Started | 19 | 30
Completed | 16 | 24
Not Completed | 3 | 6
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC | Total
Number analyzed (Participants) | 19 | 30 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.47 (10.73) | 49.17 (13.21) | 49.67 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 30 | 49
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 24 | 37
  Black or African American | 4 | 4 | 8
  Asian | 1 | 1 | 2
  Other | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 28 | 44
  Hispanic or Latino | 1 | 2 | 3
  Unknown Ethnicity | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (ypCR) Following Neoadjuvant Therapy in Breast and Axillary Lymph Nodes
Description: Percentage of patients with no histologic evidence of cancer in breast and axillary lymph nodes.
Time Frame: At the time of surgery approximately 24 to 28 weeks.
Population: 1 patient in Arm 1 was not analyzed due to inoperable, progressive disease. 2 patients in Arm 2 are missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Number analyzed (Participants) | 19 | 30
percentage of participants | 26.3 | 16.7

2. Secondary Outcome: ypCR Nodes
Description: Percentage of patients with no histologic evidence of cancer in axillary lymph nodes.
Time Frame: At the time of surgery approximately 24 to 28 weeks.
Population: 1 patient in Arm 1 was not analyzed due to inoperable, progressive disease. 2 patients in Arm 2 are missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Number analyzed (Participants) | 19 | 30
percentage of participants | 42.1 | 30.0

3. Secondary Outcome: Clinical Overall Response (cOR)(Complete and Partial) Assessed by MRI at the Completion of WP or Eribulin (Before AC)
Description: Percentage of patients with clinical complete response (no significant enhancement on MR images) or clinical partial response (at least 30% decrease in the maximal diameter of the tumor)
Time Frame: 12 weeks after initiation of study therapy
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Number analyzed (Participants) | 19 | 30
percentage of participants | 58 | 40

4. Secondary Outcome: Clinical Complete Response (ycCR) Following Neoadjuvant Therapy Assessed by Physical Exam at the Completion of Neoadjuvant Chemotherapy
Description: The number of patients with clinical complete response.
Time Frame: At approximately 24 to 28 weeks from initiation of study therapy
Population: 1 patient in Arm 1 and 3 patients in Arm 2 are missing data. The N=18 for the paclitaxel group is because analysis was done on only patients with a palpable lesion at baseline.
Measure: Number; unit: participants
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Number analyzed (Participants) | 18 | 30
participants | 8 | 10

5. Secondary Outcome: Recurrence Free Interval (RFI): The Time to Occurrence of Inoperable Progressive Disease and Local, Regional, and Distant Recurrence.
Description: The percentage of patients free from recurrence at 24 months.
Time Frame: Assessed through 24 months from randomization
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Number analyzed (Participants) | 19 | 30
percentage of patients | 83.6 [57.3 to 94.4] | 80.7 [59.6 to 91.5]

6. Secondary Outcome: 2-year Overall Survival (OS): Death From Any Cause From Time of Randomization Through 2 Years After Randomization.
Description: Percentage of patients alive at 24 months.
Time Frame: Assessed through 24 months from randomization
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Number analyzed (Participants) | 19 | 30
percentage of patients | 88.5 [61.4 to 97.0] | 92.6 [73.5 to 98.1]

7. Secondary Outcome: Adverse Events Experienced by Participants as a Measure of Toxicity.
Description: Total patients with at least 1 AE.
Time Frame: Assessed through 24 months from randomization
Population: Please refer to the AE section for more detail.
Measure: Number; unit: participants
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Number analyzed (Participants) | 19 | 30
participants | 19 | 30

ADVERSE EVENTS:
Time Frame: Emergent Adverse Events are those reported on or after the first administration and until 30 days after the last dose.
Arm/Group | Arm 1: Paclitaxel Then AC | Arm 2: Eribulin Then AC
Serious Adverse Events (participants affected / at risk) | 3/19 | 4/30
Other Adverse Events (participants affected / at risk) | 19/19 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Paclitaxel Then AC (N=19) | Arm 2: Eribulin Then AC (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Paclitaxel Then AC (N=19) | Arm 2: Eribulin Then AC (N=30)
Fatigue (General disorders) | 15 | 22
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 2
Axillary pain (General disorders) | 1 | 2
Chills (General disorders) | 1 | 2
Influenza like illness (General disorders) | 1 | 2
Mucosal inflammation (General disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 10 | 19
Constipation (Gastrointestinal disorders) | 5 | 12
Diarrhoea (Gastrointestinal disorders) | 8 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 5
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 7 | 16
Leukopenia (Blood and lymphatic system disorders) | 10 | 11
Neutropenia (Blood and lymphatic system disorders) | 10 | 11
Lymphopenia (Blood and lymphatic system disorders) | 4 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Headache (Nervous system disorders) | 5 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 5
Dysgeusia (Nervous system disorders) | 2 | 7
Dizziness (Nervous system disorders) | 3 | 2
Paraesthesia (Nervous system disorders) | 3 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 6
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 15
Aspartate aminotransferase increased (Investigations) | 1 | 7
Blood alkaline phosphatase increased (Investigations) | 1 | 5
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 4 | 6
Anxiety (Psychiatric disorders) | 1 | 6
Depression (Psychiatric disorders) | 0 | 3
Urinary tract infection (Infections and infestations) | 3 | 0
Breast pain (Reproductive system and breast disorders) | 3 | 5
Hypertension (Vascular disorders) | 1 | 4
Lacrimation increased (Eye disorders) | 2 | 1
Vision blurred (Eye disorders) | 0 | 2
Palpitations (Cardiac disorders) | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less